CLINICAL TRIAL: NCT02248623
Title: An International Multi-Centre Cohort Study of the Incidence of Anaesthesia Awareness Following Laryngoscopy and Intubation: The CONSciousness, Connectedness and IntraOperative Unresponsiveness Study (ConsCIOUS)
Brief Title: Intraoperative Anaesthesia Awareness Following Induction of Anaesthesia
Acronym: ConsCIOUS
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: University of Groningen (Other); Centre Hospitalier Régional de la Citadelle (Other); RWTH Aachen University (Other); University of Auckland, New Zealand (Other); University of Michigan (Other); University of Witten/Herdecke (Other); University College London Hospitals (Other)
Responsible Party: Sponsor
Other Study IDs: ConsCIOUS
Record Dates: First submitted 2014-09-02; First posted 2014-09-25 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Anaesthesia
Keywords: Anaesthesia; Isolated forearm test; Responsiveness; Laryngoscopy; Intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A primary aim of anaesthesia is to prevent awareness of surgery; ablation of the experience of surgery is the most secure way to prevent awareness with recall. Fortunately the incidence of awareness with recall (the patient can spontaneously remember the intraoperative event) is very rare (0.1-0.2%). However the investigators systematic review suggests that consciousness of intraoperative events may occur in approximately 37% of patients in experimental studies (as identified by the validated clinical procedure the isolated forearm test that does not require postoperative recall of the event). In this international cohort study, recruiting a minimum sample of 200 patients, the investigators will investigate the incidence of anaesthesia awareness (as identified by the isolated forearm test) following the induction of anaesthesia and before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients clinically requiring intubation will be included in this cohort.
* Patients must be able to follow the isolated forearm technique commands when awake and prior to their operation will be included in this cohort.

Exclusion Criteria:

* Contraindication to isolated forearm technique test such as unable to have tourniquet on arm for the isolated forearm technique (e.g. lymphedema or operative site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing anaesthesia requiring intubation and layngoscopy
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Incidence of isolated forearm test responsiveness following laryngoscopy and intubation | The test will occur within one minute of securing the airway (laryngoscopy and intubation).
  Following induction of anaesthesia, and securing the airway (laryngoscopy and intubation) the patient will be asked to squeeze the anaesthetist's hand as a surrogate of awareness under anaesthesia.

SECONDARY OUTCOMES:
Incidence of isolated forearm test responsiveness before laryngoscopy and intubation | The test will occur in the minute prior to securing the airway (laryngoscopy and intubation).
  Following induction of anaesthesia, and prior to securing the airway (before laryngoscopy and intubation) if safe to do so, the patient will be asked to squeeze the anaesthetist's hand as a surrogate of anaesthesia awareness.
Incidence of anaesthesia awareness with recall | Within 24 hours of the operation
  After the operation and emergence from anaesthesia, and within 24 hours of the operation, the patient will be asked, using the structured Modified Brice questionnaire, about recall of intraoperative events (anaesthesia awareness).
Patient satisfaction questionnaire | Within 24 hours of the operation and emergence from anaesthesia
  Within 24 hours of the operation and emergence from anaesthesia, the patient will be asked to complete a patient satisfaction questionnaire rating the anaesthetic care they received. This will cover the preoperative information they were given, their emergence from anaesthesia, their pain control, experience of nausea and vomiting and their general experience. They will be asked to rate their care from four options: very satisfied, satisfied, dissatisfied and very dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Sanders, MBBS PhD FRCA, Principal Investigator — University of Wisconsin, Madison
Locations (3):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - University of Wisconsin, Madison, Wisconsin
- University of Auckland, Hamilton, Waikato Region, New Zealand

REFERENCES:
- [Derived] Gaskell AL, Hight DF, Winders J, Tran G, Defresne A, Bonhomme V, Raz A, Sleigh JW, Sanders RD. Frontal alpha-delta EEG does not preclude volitional response during anaesthesia: prospective cohort study of the isolated forearm technique. Br J Anaesth. 2017 Oct 1;119(4):664-673. doi: 10.1093/bja/aex170. PMID 29121278